CLINICAL TRIAL: NCT06778096
Title: Transdiagnostic Internet Cognitive-behavior Therapy for Mixed Anxiety and Depressive Symptoms in Postnatal Women
Acronym: postnataIiCBT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre hospitalier universitaire de Sherbrooke (Unknown); Centre intégré de santé et services sociaux de la Montérégie-Centre (Unknown); Centre intégré de santé et services sociaux de la Montérégie-Ouest (Unknown); Centre intégré de santé et services sociaux de la Montérégie-Est (Unknown); Champlain Local Health Integration Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-31-2024-5238
Record Dates: First submitted 2024-12-23; First posted 2025-01-16 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Postnatal Depression
Keywords: Cognitive Behavioral Therapy; Internet; Non-guided; Transdiagnostic; Randomized clinical trial; Anxiety; Depression; Postnatal
MeSH Terms: conditions — Anxiety Disorders; Depression, Postpartum; Depression

STUDY DESIGN:
Intervention Model Description: The study design is a hybrid type 1 effectiveness-implementation study. The clinical trial is a two-arm parallel group multicentre pragmatic superiority RCT, with allocation at the level of the individual. This study is an adaptation that will follow the original postnatal anxiety and depression iCBT program clinical trial (Loughnan et al., 2019). The proposed trial is congruent with CONSORT recommendations for RCTs and nonpharmacological treatments. The postnatal iCBT program will be offered to participants in the TAU condition at the end of the four-week follow-up (delayed-intervention).
Masking Description: Participants and research coordinator will not be blinded in regard to the participants group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The postnatal anxiety and depression iCBTprogram + TAU (Experimental): Women will have access to the postnatal iCBT program (self-directed) and will have to complete the program over six weeks. They still can have contacts with the healthcare system.
  Interventions: Behavioral: Postnatal anxiety and depression iCBTprogram
- Treatment-as-usual (No Intervention): No restrictions will be imposed regarding usual care. To reflect heterogeneity of health seeking behaviour and mental health practices for anxiety and depressive symptoms in the community during the postpartum period, participants will not be constrained to a prespecified usual care treatment for external validity or have contacts with the healthcare system. Data will be collected on throughout the trial. This group will have a delayed access to the program after they complete their four-week follow-up questionnaire.

INTERVENTIONS:
Behavioral: Postnatal anxiety and depression iCBTprogram — The overarching goal of this stand-alone program is to introduce women to CBT skills to help manage symptoms of anxiety and depression, such as psychoeducation, cognitive restructuring and problem solving, behavioural activation, graded exposure and relapse prevention. Each lesson is accompanied by practical homework and resources (e.g., medication during breastfeeding, attachment and bonding, information for entourage, sleep, self-care, intrusive thought, problem solving), and is built to be easily generalizable to a broad range of women. The three lessons must be completed within a 6-week period, with up to two weeks to complete each lesson. Participants will be notified of new lessons available via email and text message reminders. There is a 5-day lockout between lessons stopping the participants to complete the next session once a session is completed to ensure that the sessions are completed over multiple weeks to allow for revision and practice.
  Other Names: Postnatal iCBT
  Arms: The postnatal anxiety and depression iCBTprogram + TAU

SUMMARY:
This research project aims to examine the acceptability and efficacy of a French-Canadian adaptation of a postnatal anxiety and depression program. The main question it aims to answer is:

[1] When the adapted postnatal Internet-delivered cognitive behavioral therapy (iCBT) is added to treatment as usual (TAU) in community-based care for women with anxiety and depressive symptoms, is the iCBT+TAU condition more effective to reduce symptoms than TAU alone?

Participants will:

postnatal iCBT group -> Answer questionnaires before, after (week 6) and 4 weeks after the intervention (week 10); do the 6-week non-guided iCBT program for anxiety and depressive symptoms during the postnatal period.

Waitlist, TAU group -> Answer questionnaires at enrolment, at week 6 and week 10. Participants will have access to the intervention after they complete their last questionnaires.

DETAILED DESCRIPTION:
Background. Nearly 20% of women will be confronted with anxiety or depressive disorders during the perinatal period and this may lead to adverse outcomes for both mother and child. Cognitive behavioural therapy (CBT) is the psychological intervention with the most empirical support for the clinical management of anxiety and depressive disorders. Depression and anxiety frequently occur in women during the perinatal period, and there is growing evidence that internet-delivered CBT (iCBT) could be an acceptable and effective intervention. ThisWayUp iCBT Virtual Clinic in Australia has developed a program for postnatal anxiety and depression. As part of a Québec-Ontario collaboration, this research protocol aims to examine the acceptability and efficacy of a French-Canadian adaptation of the postnatal anxiety and depression program. Methods/Design. The investigators propose to conduct a hybrid type 1 randomized clinical trial and implementation study to replicate the findings of the trial conducted in Australia as well as explore barriers and facilitators to potential large-scale implementation. Treatment and control groups. a) adapted postnatal depression and anxiety iCBT program (3 lessons to complete in six weeks) added to treatment-as-usual (TAU); b) TAU. Participants will include women with possible postnatal depression or anxiety as per the Generalized Anxiety Disorder-7 (GAD-7) or the Edinburgh Postnatal Depression Scale (EPDS). The primary outcome measures will be the GAD-7 and the EPDS. Secondary outcome measures will comprise self-reported instruments to evaluate mother-child experience, postnatal depression, psychological distress, suicidality risk, quality of life, treatment satisfaction and service utilization. Statistical analysis. Statistical analysis will follow intent-to-treat principles. A mixed model regression approach will be used to account for between- and within-subject variations in the analysis of the longitudinal effects of iCBT compared to TAU intervention. Moderation analyses will be performed for three sets of moderators: clinical characteristics, previous treatments and sociodemographic characteristics. Additionally, treatment effect sizes will be calculated with Cohen's d. Discussion. The study will deliver important data of efficacy and acceptability to patients, clinicians, and decision-makers to inform the scaling-up of the postnatal iCBT intervention. The benefits to patients could include timely access to services, improved remission rates and health-related quality of life, better long-term outcomes; and to the healthcare system, policy and decision-makers: improved efficiency, optimization of resources, and this to meet the perinatal women and child needs equitably.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Being within 12 months postpartum
* Fluent in spoken and written French
* Self-reported clinical score ≥10 for anxiety and/or depressive symptoms based on the Generalised Anxiety Disorder-7 (GAD-7) and the Edinburgh Postnatal Depression Scale 10-item scale (EPDS)
* Access to a computer/tablet and internet connection
* Agreement to share primary provider contact information

Exclusion Criteria:

* Self-reported diagnosis of schizophrenia or bipolar disorder
* Current substance abuse or dependence
* Current use of benzodiazepines
* Beginning psychological therapy (< 4 weeks ago) or medication (< 8 weeks ago) for depression/anxiety
* Severe depression (EPDS score ≥ 23) or active suicidal intentions (EPDS question 10 = 3, yes quite often)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (French) | Week 0, Week 6, Week 10
  Used to evaluate postpartum depression. 10 items, 0 to 3 Likert scale, retrospective on the past 7 days. The score varies between 0 and 30, with a higher score indicating more severe symptoms.
Generalised Anxiety Disorder-7 (French) | Week 0, Week 6, Week 10
  Used to evaluate the severity of anxiety symptoms. 7 items, 0 to 3 Likert scale, retrospective on the past 14 days. The score varies between 0 and 21, with a higher score indicating more severe symptoms.

SECONDARY OUTCOMES:
Kessler Psychological Distress Scale - 10 items (French) | Week 0, before each program lesson (intervention group) Week 6, Week 10
  Used to evaluate psychological distress. 10 items, 1 to 5 Likert scale, retrospective on the past 14 days. The score varies between 10 and 50, with a higher score indicating more psychological distress.
Assessment of Quality of Life - 6 dimensions (French) | Week 0, week 6 and week 10
  20-item self-administered health-related quality of life tool, retrospective over the past week, to be rated on Likert scales with varying number of levels. It assesses six dimensions: independent living, mental health, coping, relationships, pain, senses. Response options for each item range from 4-6 levels. Scores on each domain and a total score can be derived. Standardized scores range from 0 to 100 where higher scores indicate less quality of life impairment.
Maternal Postnatal Attachment Scale (French) | Week 0, Week 6 and Week 10
  19-item self-report questionnaire to assess the affective aspect of mother-infant bonding over the past 2 weeks. It is based on three subscales: absence of hostility, pleasure in interaction and quality of attachment. The score varies between 19 and 95; lower scores indicate more problematic responses.

OTHER OUTCOMES:
Client Satisfaction Questionnaire (8-item French version) | Week 6
  Tool for evaluating client's satisfaction with a service. It consists of eight items to be evaluated on a 4-point Likert scale. The score varies between 8 and 32, with a higher score indicating greater satisfaction.
System Usability Scale | Week 6
  It measures the efficiency of a system as well as its effectiveness perceived by users and also their satisfaction. The scale goes from 0 to 100, where a higher score indicates higher usability.
Past health service utilization | Week 0 (baseline, retrospective on the past 3 months), Week 6 (post-treatment, retrospective on the past 6 weeks), Week 10 (follow-up, retrospective on the past 4 weeks)
  Visits with health professionals (number, type of professionnals), previous psychotherapy for anxiety or depression (yes/no, additional true/false questions about the psychotherapy they received), medication (name). These data will be used for descriptive analysis or control variables.

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Roberge, PhD, Principal Investigator — Université de Sherbrooke; Helen-Maria Vasiliadis, PhD, Principal Investigator — Université de Sherbrooke
Locations (4):
- Canada (4):
  - Centre intégré de santé et services sociaux de la Montérégie-Ouest, Châteauguay, Quebec
  - Centre intégré de santé et services sociaux de la Montérégie-Est, Greenfield Park, Quebec
  - Centre intégré de santé et services sociaux de la Montérégie-Centre, Longueuil, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No
The datasets generated during the current study will not be publicly available due to ethics committee regulations, but will be available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Loughnan SA, Butler C, Sie AA, Grierson AB, Chen AZ, Hobbs MJ, Joubert AE, Haskelberg H, Mahoney A, Holt C, Gemmill AW, Milgrom J, Austin MP, Andrews G, Newby JM. A randomised controlled trial of 'MUMentum postnatal': Internet-delivered cognitive behavioural therapy for anxiety and depression in postpartum women. Behav Res Ther. 2019 May;116:94-103. doi: 10.1016/j.brat.2019.03.001. Epub 2019 Mar 8. No abstract available. PMID 30877878
- [Derived] Roberge P, Vasiliadis HM, Chapdelaine A, Battista MC, Beaulieu MC, Chomienne MH, Cumyn A, Drapeau M, Durand C, Girard A, Gosselin D, Grenier J, Hardy I, Hudon C, Koszycki D, Labelle R, Lesage A, Lussier MT, Mahoney A, Provencher MD, Shiner CT. Transdiagnostic internet cognitive behavioural therapy for anxiety and depressive symptoms in postnatal women: protocol of a randomized controlled trial. BMC Psychiatry. 2025 Mar 13;25(1):237. doi: 10.1186/s12888-025-06636-3. PMID 40075340